CLINICAL TRIAL: NCT07063290
Title: COMBO Endoscopy Oropharyngeal Airway in Sedated Fiberoptic Bronchoscopy for Patients: A Simon Two-Stage Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, chair of Anesthesiology Department, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025B0779
Record Dates: First submitted 2025-06-29; First posted 2025-07-14 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Infection; Pulmonary Nodule; Endotracheal Tumour; Bronchiectasis
Keywords: the COMBO Endoscopy Oropharyngeal Airway; fiberoptic bronchoscopy; hypoxia
MeSH Terms: conditions — Bronchiectasis; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the COMBO Endoscopy Oropharyngeal Airway Group (Other): In this group, patients use the COMBO Endoscopy Oropharyngeal Airway for oxygenation.
  Interventions: Device: the COMBO Endoscopy Oropharyngeal Airway

INTERVENTIONS:
Device: the COMBO Endoscopy Oropharyngeal Airway — Using the COMBO Endoscopy Oropharyngeal Airway for oxygenation.

SUMMARY:
Hypoxia represents the prevailing adverse occurrence during the sedation of patients undergoing fiberoptic bronchoscopy with propofol. A recent innovation in this domain is the COMBO Endoscopy Oropharyngeal Airway-a multifaceted device that encompasses capnography monitoring, bite block , oxygenation support, and oropharyngeal airway management. This device has been purposefully designed to cater to the unique requirements of endoscopic procedures. The principal objective of our randomized study is to assess the efficacy and safety of the COMBO Endoscopy Oropharyngeal Airway reduce the incidence of hypoxia on patients undergoing fiberoptic bronchoscopy under propofol sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18≤ Age ≤60.·Patients undergoing fiberoptic bronchoscopy.
* Patients have signed the informed consent form.
* The ASA classification ranges from I to II.
* The estimated duration of the procedure does not exceed 45 minutes.

Exclusion Criteria:

* Patients with contraindications to oropharyngeal airway ventilation, such as coagulation disorders, predisposition to oral/nasal bleeding, mucosal damage, or anatomical obstructions hindering oropharyngeal airway placement.
* Patients diagnosed with acute exacerbation of chronic obstructive pulmonary disease (COPD) or those currently suffering from other acute/chronic pulmonary conditions requiring long-term or intermittent oxygen therapy.
* Patients with preoperative SpO₂ < 95% while breathing air.
* Patients with BMI < 18.5 or BMI > 30.
* Patients with upper respiratory tract infections (oral, nasal, or pharyngeal).
* Patients at risk of aspiration.
* Patients with fever (core temperature > 37.5°C).
* Patients with severe cardiac insufficiency (< 4 METs).
* Patients with severe renal insufficiency requiring preoperative dialysis.
* Patients with a confirmed diagnosis of hepatic insufficiency.
* Patients with increased intracranial pressure.
* Patients with hypersensitivity to sedatives like propofol or medical equipment such as adhesive tape.
* Patients with a history of drug abuse and/or alcoholism within the two years preceding the commencement of the screening period (defined as drinking more than three standard alcoholic beverages daily, roughly equivalent to 10g of alcohol or 50g of Chinese Baijiu).
* Patients with a history of mental and neurological disorders, including but not limited to depression, severe central nervous system depression, Parkinson's disease, basal ganglia lesions, schizophrenia, epilepsy, Alzheimer's disease, and myasthenia gravis.
* Patients currently participating in other clinical trials.
* Patients deemed ineligible for participation in this clinical trial by the researchers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia（75% ≤ SpO2 < 90% for <60 s） | Patients are continuously monitored from the beginning of anesthesia induction until exiting the PACU (Post-Anesthesia Care Unit).

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression（90% ≤ SpO2 < 95%） | Patients are continuously monitored from the beginning of anesthesia induction until exiting the PACU (Post-Anesthesia Care Unit).
The incidence of severe hypoxia（SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s） | Patients are continuously monitored from the beginning of anesthesia induction until exiting the PACU (Post-Anesthesia Care Unit).

OTHER OUTCOMES:
The incidence of other adverse events | Patients are continuously monitored from the beginning of anesthesia induction until exiting the PACU (Post-Anesthesia Care Unit).
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital, Zhejiang University School Of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided